CLINICAL TRIAL: NCT06416241
Title: Intravitreal Aflibercept for Macular Edema Due to Central Retinal Vein Occlusion
Acronym: INTRAMED-CRVO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Irini Chatziralli, Associate Professor in Ophthalmology, National and Kapodistrian University of Athens
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 699/2019
Record Dates: First submitted 2024-05-08; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Retinal Vein Occlusion; Vascular Occlusive Disease
Keywords: optical coherence tomography angiography; aflibercept; retinal vein occlusion; biomarkers
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — aflibercept; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Eylea 2.0mg/0.05ml (Other)
  Interventions: Drug: EYLEA 2 MG in 0.05 ML Injection

INTERVENTIONS:
Drug: EYLEA 2 MG in 0.05 ML Injection — Intravitreal injection

SUMMARY:
Central retinal vein occlusion (CRVO) is a common retinal vascular disorder, occurring when there is a blockage to the main blood vessel that transports blood away from the retina. CRVO may cause visual impairment, especially due to macular edema (swelling of the macula due to fluid accumulation) and macular non-perfusion.

Aflibercept has been found to improve visual acuity and reduce macular thickness in pivotal trials.

The purpose of this study was to evaluate the efficacy and safety of intravitreal aflibercept in real-world, using a patient-fitted treatment regimen. Additionally, imaging parameters have been assessed before and after treatment with intravitreal aflibercept.

ELIGIBILITY:
Inclusion Criteria:

* Treatment naive center-involved macular edema secondary to CRVO for no longer than 3 months.
* Patients >18 years of age, who are diagnosed with macular edema secondary to CRVO who are scheduled to be treated with intravitreal aflibercept in real-life conditions
* BCVA of Snellen of 20/40 to 20/200 in the study eye

Exclusion Criteria:

* Previous PRP or macular laser photocoagulation in the study eye.
* Any prior ocular treatment in the study eye for macular edema secondary to CRVO.
* Prior systemic anti-VEGF or corticosteroid therapy, within the last 3 months before enrollment to the study.
* Any active or previous inflammation, ocular trauma
* Uncontrolled glaucoma (IOP>30 mmHg)

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Change in visual acuity as measured using ETDRS charts | 5 years
Change in retinal thickness as measured in μm using spectral domain optical coherence tomography | 5 years

SECONDARY OUTCOMES:
Change in microvascular parameters in OCT angiography (vessel density, FAZ area) | 2 years
Complications | 5 years
Change in endothelial dysfunctionafter aflibercept treatment, as measured by the perfused boundary region sublingual 5-25 μm | 6 months